CLINICAL TRIAL: NCT06181669
Title: Pneumonia Direct Pilot
Acronym: PDP
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00113767; 5UM1AI104681 (NIH)
Record Dates: First submitted 2023-11-20; First posted 2023-12-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pneumonia, Bacterial; Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endotracheal suctioning (ETS) fluid samples, Bronchoalveolar (BAL) lavage fluid, bacterial isolates, whole blood, serum, and plasma will be sent to a central research laboratory for host- and pathogen-diagnostic testing. Back up samples will stored at the ARLG Laboratory Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Standard of Care: There are no interventions in this study. Standard of care activities will be captured in the eCRF and samples will be collected and tested. Results will not be returned to the sites or participants.
  Interventions: Diagnostic Test: Pathogen and Host Directed testing

INTERVENTIONS:
Diagnostic Test: Pathogen and Host Directed testing — This study will compare up to 6 pathogen-directed tests and 3 host biomarker tests. Pathogen-directed tests detect and identify the most common causes of bacterial pneumonia, while host biomarker tests assess the host's immune response to infection. Testing will occur at various testing centers.
  Evaluable participant specimens will be sent to a central laboratory for distribution to the testing centers that will perform the index testing. Testing centers will be blinded to whether the samples were collected at baseline or clinical change. Further, each testing center will prepare and test the specimens according to documented procedures, then transfer the testing results to the ARLG Statistics and Data Management Center for analysis. Neither the study sites, participants, nor adjudicators will receive the results from the index testing. After the study, untested aliquots of specimens will be stored in the ARLG Physical Biorepository.
  Other Names: Respiratory Pathogen ID/AMR Enrichment Panel (Illumina); Metagenomic Next Generation Sequencing (Illumina); T2 Bacteria Panel (T2 Biosystems); T2 Resistance Panel (T2 Biosystems); Procalcitonin (Abbott); TriVerity host (Inflammatix); Host gene expression; FilmArray Pneumonia Panel (BioFire)

SUMMARY:
The Pneumonia Direct Pilot study is designed to assess whether combining molecular diagnostics for bacteria and AMR markers with host-response profiling improves agreement and predictive value for the diagnosis of VAP versus an adjudicated clinical reference standard. The feasibility design is intended to inform future interventional studies that will investigate the clinical impact of combined pathogen- and host-directed testing approaches.

DETAILED DESCRIPTION:
This is a prospective, observational, diagnostic, feasibility study to determine the accuracy of pathogen- and host-directed testing for the diagnosis of VAP. Newly intubated adult patients admitted to the ICU will be assessed for eligibility around the time of intubation according to the inclusion/exclusion criteria. Screening and consent can occur any time within 48 hours of a patient being intubated. Between 48 and 60 hours after intubation, eligible participants will have blood drawn and dedicated research aliquots from SOC ETS samples retrieved. The dedicated research aliquots from SOC ETS samples will be obtained simultaneously with routine sampling for microbiologic testing or, when this is not possible, during routine suctioning as a part of standard airway care. Collection of other clinical data may occur 24 to 72 hours after intubation.

Participants will be followed daily for a clinical change for up to 14 days from the time of intubation. Clinical change is defined as a clinical suspicion of new-onset VAP that prompts the collection of lower respiratory tract secretions for routine microbiologic testing and initiation, continuation, or modification of antibiotic therapy for a pneumonia indication.

Participants who experience a clinical change will have additional blood samples drawn and dedicated aliquots of the sample retrieved from standard-of-care ETS procedures. Additionally, if available, leftover bronchoalveolar lavage (BAL) will be reclaimed, and respiratory and blood bacterial isolates will be obtained from SOC cultures. Participants will be followed through the diagnosis of clinical change and finalization of all local microbiological and radiological results obtained as a part of usual care. Clinical data will be recorded through medical record review.

Participants who do not experience a clinical change will be followed through extubation, ICU discharge, death, or for up to 14 days after intubation - whichever comes first. Participants who do not have a clinical change will not undergo additional sample collection.

Clinical change events will be used to assess whether the participant meets the clinical case definition (FDA criteria) for VAP: VAP-positive (VAP+) or VAP-negative (VAP-) categories will be obtained by an algorithm linked to the eCRF data. The VAP clinical case definition will be adjudicated against the participants' clinical data and microbiological evidence and the certainty of the VAP diagnosis will be classified as follows: Prove, Probable, Possible VAP, or No VAP. Every participant with a clinical change will be assessed for the presence of an extrapulmonary infection. Extrapulmonary infection will be classified as follows: Proven, Possible, or No Infection.

Evaluable participant specimens will be sent to a central laboratory for distribution to the testing centers that will perform the index testing. This study will compare pathogen-directed tests and host biomarker tests. Pathogen-directed tests detect and identify the most common causes of bacterial pneumonia, while host biomarker tests assess the host's immune response to infection. Testing centers will be blinded to whether the samples were collected at baseline or clinical change. Neither the study sites, participants, nor adjudicators will receive the results from the index testing.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥18 years old
2. Are newly intubated for less than 48 hours and for reasons other than suspected bacterial pneumonia or suspected acute bacterial infection
3. Are expected to require intubation for at least 48 hours, per the discretion of the treating clinician
4. Are able to provide protocol-accepted consent (legally authorized representative [LAR] is acceptable)
5. Are expected to live long enough to receive a VAP diagnosis, at the discretion of the treating clinician
6. Are able to provide study-required biological samples

Exclusion Criteria:

1. Have a witnessed or suspected aspiration event prompting the need for current, new intubation
2. Have known active lung cancer or metastatic disease to a lung
3. Received a lung transplant
4. Have cystic fibrosis
5. Are receiving comfort care
6. Are receiving antibiotic treatment for suspected or proven active acute bacterial infection (eg, pneumonia, tracheobronchitis, sepsis)
7. Have a current or within-the-last-30-days diagnosis of active bacterial pneumonia
8. Were previously enrolled in this trial
9. Require long-term ventilator support
10. Have a tracheostomy tube in place
11. Are currently participating in an interventional drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated adult patients (≥18 years of age) admitted to the ICU will be assessed for eligibility around the time of intubation according to the inclusion/exclusion criteria. Screening and consent may occur at any time within 48 hours of patients being intubated. The target sample size is 250 participants in order to observe approximately 30 clinical VAP-positive cases. Vulnerable patients, including women and minorities, will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of participants with positive results on the Respiratory Pathogen ID/AMR Enrichment Panel (Illumina) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the Metagenomic Next Generation Sequencing (Illumina) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the T2 Bacteria Panel (T2 Biosystems) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the T2 Resistance Panel (T2 Biosystems) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the Procalcitonin (Abbott) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the TriVerity host (Inflammatix) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the Host gene expression | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
The number of participants with positive results on the FilmArray Pneumonia Panel (BioFire) | Through study completion, or up to 18 months, whichever comes first
  This study will compare the results (positive, negative, or no result) of each index test.
Number of participants with a clinical diagnosis of VAP at the time of clinical change | day 15
  * Clinical diagnosis of VAP is defined as new findings in each category of signs and imaging
    o At least one of the following signs of inflammation: Fever >=38 °C or =35 °C Leukocytosis (white blood cell count ≥12K/mm3 or ≤4K/mm3) >15% immature neutrophils (bands) AND
    * signs of respiratory worsening. AND
    * New or progressive changes suggestive of bacterial pneumonia from imaging: infiltrate, consolidation, and/or cavitation
  * Clinical change is defined as a clinical suspicion of new onset VAP that prompts collection of lower respiratory tract secretions for routine microbiologic testing and initiation or continuation of empiric antibiotic therapy for a pneumonia indication.

SECONDARY OUTCOMES:
Number of participants with an adjudicated diagnosis of of proven, probable, possible, or no VAP at the time of clinical change utilizing clinical and microbiological information | through extubation, ICU discharge, death, or for up to 14 days after intubation - whichever comes first
  - clinical information collected from participants with a clinical change will be reviewed to discern the presence of signs and symptoms of VAP as well as evidence of extrapulmonary infection. Cases of suspected VAP and extra-pulmonary infection will then be classified as proven, probable/possible or no infection using expert adjudication and standardized definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly E Hanson, MD, MHS, Principal Investigator — University of Utah
Locations (4):
- United States (4):
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell (William Beaumont), Royal Oak, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
During the analysis process, diagnostic companies will support the testing of some specimens and will provide the resulting data back to the Duke Clinical Research Institute.
  Once clinical and laboratory data have been analyzed and the primary manuscript has been published, investigators may apply to the Antibacterial Resistance Leadership Group (ARLG) for use of data. Continued regulatory oversight, Data Use Agreements, and Material Transfer agreements may apply.
Supporting Information: Study Protocol
Time Frame: Once the primary manuscript has been published
Access Criteria: Application to the ARLG for use

REFERENCES:
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Safdar N, Dezfulian C, Collard HR, Saint S. Clinical and economic consequences of ventilator-associated pneumonia: a systematic review. Crit Care Med. 2005 Oct;33(10):2184-93. doi: 10.1097/01.ccm.0000181731.53912.d9. PMID 16215368
- [Background] Kuti EL, Patel AA, Coleman CI. Impact of inappropriate antibiotic therapy on mortality in patients with ventilator-associated pneumonia and blood stream infection: a meta-analysis. J Crit Care. 2008 Mar;23(1):91-100. doi: 10.1016/j.jcrc.2007.08.007. PMID 18359426
- [Background] Nussenblatt V, Avdic E, Berenholtz S, Daugherty E, Hadhazy E, Lipsett PA, Maragakis LL, Perl TM, Speck K, Swoboda SM, Ziai W, Cosgrove SE. Ventilator-associated pneumonia: overdiagnosis and treatment are common in medical and surgical intensive care units. Infect Control Hosp Epidemiol. 2014 Mar;35(3):278-84. doi: 10.1086/675279. Epub 2014 Feb 3. PMID 24521594
- [Background] Klompas M. Does this patient have ventilator-associated pneumonia? JAMA. 2007 Apr 11;297(14):1583-93. doi: 10.1001/jama.297.14.1583. PMID 17426278
- [Background] Khan S, Liu J, Xue M. Transmission of SARS-CoV-2, Required Developments in Research and Associated Public Health Concerns. Front Med (Lausanne). 2020 Jun 9;7:310. doi: 10.3389/fmed.2020.00310. eCollection 2020. PMID 32582747
- [Background] Murphy CN, Fowler R, Balada-Llasat JM, Carroll A, Stone H, Akerele O, Buchan B, Windham S, Hopp A, Ronen S, Relich RF, Buckner R, Warren DA, Humphries R, Campeau S, Huse H, Chandrasekaran S, Leber A, Everhart K, Harrington A, Kwong C, Bonwit A, Dien Bard J, Naccache S, Zimmerman C, Jones B, Rindlisbacher C, Buccambuso M, Clark A, Rogatcheva M, Graue C, Bourzac KM. Multicenter Evaluation of the BioFire FilmArray Pneumonia/Pneumonia Plus Panel for Detection and Quantification of Agents of Lower Respiratory Tract Infection. J Clin Microbiol. 2020 Jun 24;58(7):e00128-20. doi: 10.1128/JCM.00128-20. Print 2020 Jun 24. PMID 32350043
- [Background] Charalampous T, Alcolea-Medina A, Snell LB, Williams TGS, Batra R, Alder C, Telatin A, Camporota L, Meadows CIS, Wyncoll D, Barrett NA, Hemsley CJ, Bryan L, Newsholme W, Boyd SE, Green A, Mahadeva U, Patel A, Cliff PR, Page AJ, O'Grady J, Edgeworth JD. Evaluating the potential for respiratory metagenomics to improve treatment of secondary infection and detection of nosocomial transmission on expanded COVID-19 intensive care units. Genome Med. 2021 Nov 17;13(1):182. doi: 10.1186/s13073-021-00991-y. PMID 34784976
- [Background] Gaston DC, Miller HB, Fissel JA, Jacobs E, Gough E, Wu J, Klein EY, Carroll KC, Simner PJ. Evaluation of Metagenomic and Targeted Next-Generation Sequencing Workflows for Detection of Respiratory Pathogens from Bronchoalveolar Lavage Fluid Specimens. J Clin Microbiol. 2022 Jul 20;60(7):e0052622. doi: 10.1128/jcm.00526-22. Epub 2022 Jun 13. PMID 35695488
- [Background] Sotillo-Diaz JC, Bermejo-Lopez E, Garcia-Olivares P, Peral-Gutierrez JA, Sancho-Gonzalez M, Guerrero-Sanz JE. [Role of plasma procalcitonin in the diagnosis of ventilator-associated pneumonia: systematic review and metaanalysis]. Med Intensiva. 2014 Aug-Sep;38(6):337-46. doi: 10.1016/j.medin.2013.07.001. Epub 2013 Sep 12. Spanish. PMID 24035696
- [Background] Kostaki A, Wacker JW, Safarika A, Solomonidi N, Katsaros K, Giannikopoulos G, Koutelidakis IM, Hogan CA, Uhle F, Liesenfeld O, Sweeney TE, Giamarellos-Bourboulis EJ. A 29-MRNA HOST RESPONSE WHOLE-BLOOD SIGNATURE IMPROVES PREDICTION OF 28-DAY MORTALITY AND 7-DAY INTENSIVE CARE UNIT CARE IN ADULTS PRESENTING TO THE EMERGENCY DEPARTMENT WITH SUSPECTED ACUTE INFECTION AND/OR SEPSIS. Shock. 2022 Sep 1;58(3):224-230. doi: 10.1097/SHK.0000000000001970. Epub 2022 Aug 26. PMID 36125356
- [Background] Langelier C, Kalantar KL, Moazed F, Wilson MR, Crawford ED, Deiss T, Belzer A, Bolourchi S, Caldera S, Fung M, Jauregui A, Malcolm K, Lyden A, Khan L, Vessel K, Quan J, Zinter M, Chiu CY, Chow ED, Wilson J, Miller S, Matthay MA, Pollard KS, Christenson S, Calfee CS, DeRisi JL. Integrating host response and unbiased microbe detection for lower respiratory tract infection diagnosis in critically ill adults. Proc Natl Acad Sci U S A. 2018 Dec 26;115(52):E12353-E12362. doi: 10.1073/pnas.1809700115. Epub 2018 Nov 27. PMID 30482864
- [Background] Kalantar KL, Neyton L, Abdelghany M, Mick E, Jauregui A, Caldera S, Serpa PH, Ghale R, Albright J, Sarma A, Tsitsiklis A, Leligdowicz A, Christenson SA, Liu K, Kangelaris KN, Hendrickson C, Sinha P, Gomez A, Neff N, Pisco A, Doernberg SB, Derisi JL, Matthay MA, Calfee CS, Langelier CR. Integrated host-microbe plasma metagenomics for sepsis diagnosis in a prospective cohort of critically ill adults. Nat Microbiol. 2022 Nov;7(11):1805-1816. doi: 10.1038/s41564-022-01237-2. Epub 2022 Oct 20. PMID 36266337
- [Background] Bergin SP, Coles A, Calvert SB, Farley J, Powers JH, Zervos MJ, Sims M, Kollef MH, Durkin MJ, Kabchi BA, Donnelly HK, Bardossy AC, Greenshields C, Rubin D, Sun JL, Chiswell K, Santiago J, Gu P, Tenaerts P, Fowler VG Jr, Holland TL. PROPHETIC: Prospective Identification of Pneumonia in Hospitalized Patients in the ICU. Chest. 2020 Dec;158(6):2370-2380. doi: 10.1016/j.chest.2020.06.034. Epub 2020 Jun 29. PMID 32615191
- [Background] Bergin SP, Calvert SB, Farley J, Sun JL, Chiswell K, Dieperink W, Kluytmans J, Lopez-Delgado JC, Leon-Lopez R, Zervos MJ, Kollef MH, Sims M, Kabchi BA, Rubin D, Santiago J, Natarajan M, Tenaerts P, Fowler VG, Holland TL, Bonten MJ, Hullegie SJ. PROPHETIC EU: Prospective Identification of Pneumonia in Hospitalized Patients in the Intensive Care Unit in European and United States Cohorts. Open Forum Infect Dis. 2022 May 9;9(7):ofac231. doi: 10.1093/ofid/ofac231. eCollection 2022 Jul. PMID 35836748
- [Background] Corneli A, Calvert SB, Powers JH 3rd, Swezey T, Collyar D, Perry B, Farley JJ, Santiago J, Donnelly HK, De Anda C, Blanchard K, Fowler VG Jr, Holland TL. Consensus on Language for Advance Informed Consent in Health Care-Associated Pneumonia Clinical Trials Using a Delphi Process. JAMA Netw Open. 2020 May 1;3(5):e205435. doi: 10.1001/jamanetworkopen.2020.5435. PMID 32442291
- See also: The BioFire® FilmArray®Pneumonia (PN) Panel. BioFire Diagnostics. 2023. — https://www.biofiredx.com/products/the-filmarray-panels/filmarray-pneumonia
- See also: FDA. Hospital-Acquired Bacterial Pneumonia and Ventilator-Associated Bacterial Pneumonia: Developing Drugs for Treatment Guidance for Industry. Accessed October 20, 2022. — https://www.fda.gov/media/79516/download